CLINICAL TRIAL: NCT02034318
Title: Fatigue and Cardiac Sympathetic Denervation in Parkinson Disease
Acronym: Fatigue
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Carlos Singer, Carlos Singer, MD, University of Miami
Other Study IDs: 20090004
Record Dates: First submitted 2013-12-11; First posted 2014-01-13 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: Fatigue; Cardiac Sympathetic Denervation; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research study is to learn about a possible association between cardiac denervation (the breaking down of nerves in the heart) and the development of fatigue in Parkinson's disease (PD).

DETAILED DESCRIPTION:
This investigator-initiated study is meant to determine whether a correlation exists between cardiac denervation (as assessed by 123I-mIBG scans) and subjective ratings of fatigue in patients with Parkinson disease. Subjects will be recruited from the Movement Disorder section of the department of Neurology. Subjects fulfilling inclusion/exclusion criteria will undergo testing to exclude confounding factors such as depression or sleep dysfunction. Subjects will also complete several validated measures of fatigue. These measures will be correlated to a calculated ratio obtained from an 123I-mIBG scan to provide an indication of the relative denervation present in the subject. These findings will serve as pilot data for a larger prospective study exploring this topic.

Patients who are found to have possible signs of depression based on the depression ratings scales performed during the study will be provided with a referral to a mental health specialist for further evaluation and treatment. Patients who endorse thoughts of suicide or homicide will be referred to the Jackson Memorial Mental Health Crisis Intervention Center for acute evaluation.

The radiopharmaceutical 123-I-mIBG has been approved for assessing sympathetic activity in neuroendocrine tumors and is currently undergoing investigation in the study of sympathetic innervations of the heart in heart failure and a variety of other electrophysiologic abnormalities of the heart, in which sympathetic innervations may be playing a role. The subject will be exposed to small doses of radiation during the course of the scan. Nuclear medicine has been used for more than five decades, and there are no known long-term adverse effects from such low-dose exposure. Allergic reactions to radiopharmaceuticals may occur but are extremely rare and are usually mild. This risk will be minimized by excluding individuals with previous allergic reactions to iodine. Injection of the radiotracer may cause slight pain and redness which should rapidly resolve. Some medications may have to be stopped a few hours before the 123-I-mIBG scan is performed.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Parkinson's disease within the past 5 years
* Have mild to moderate Parkinson's disease (H&Y Stage ≤ 3)

Exclusion Criteria:

* Are currently pregnant or lactating
* Fulfill DSM IV TR criteria for major depression or dysthymia
* Fulfill DSM criteria for generalized anxiety disorder or panic disorder
* Are currently taking a medication known to affect 123I-mIBG uptake (See Appendix 1)
* Have a history of previous relevant cardiac disease, or any clinically significant abnormalities on routine chest radiography, electrocardiography, or cardiac ultrasonography
* Have active lung disease, including asthma, COPD, or pneumonia
* Have diabetes mellitus
* Have congestive heart failure
* Have an active systemic infection
* History of allergic reaction to radionuclide agent or have allergy to iodine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly/aged Outpatients
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2009-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Comparison of cardiac uptake with fatigue severity score | six weeks
  The purpose of this research study is to learn about a possible association between cardiac denervation (the breaking down of nerves in the heart) and the development of fatigue in Parkinson's disease (PD).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States